CLINICAL TRIAL: NCT06067490
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose (SAD) Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, andImmunogenicity of RC1416 Injection Via Subcutaneous Administration in Healthy Adult Volunteers.
Brief Title: A Phase I Study of RC1416 Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing RegeneCore Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NJRJK-RC1416-Ia
Record Dates: First submitted 2023-09-12; First posted 2023-10-05 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RC1416 (Experimental): RC1416(SAD),single ascending (25mg-600mg) of RC1416 by subcutaneous injection
  Interventions: Drug: RC1416(SAD)
- Placebo (Placebo Comparator): Placebo(SAD), Each subjects will receive the placebo once by subcutaneous injection.
  Interventions: Drug: Placebo(SAD)

INTERVENTIONS:
Drug: RC1416(SAD) — RC1416(SAD),there are six doses(25mg-600mg) in this part. Each subjects will receive the drug once by subcutaneous injection.
  Other Names: RC1416
  Arms: RC1416
Drug: Placebo(SAD) — Placebo(SAD), Each subjects will receive the placebo once by subcutaneous injection.
  Other Names: RC1416 Placebo
  Arms: Placebo

SUMMARY:
This is a phase I study to evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of RC1416 injection via Subcutaneous Administration in Healthy Adult Volunteers.

DETAILED DESCRIPTION:
RC1416 is a bispecific homodimer nanobody .It is being developed by Nanjing RegeneCore Biotech Co., Ltd. as a potential therapy for asthma. A total 48 healthy adult subjects will be enrolled in six groups to access the safety and tolerability of single subcutaneous injection of RC1416 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 50 years(including the boundary value)，Chinese.
* Male Weight of 50 kg to 90 kg，femal weight of 40kg to 90kg, and BMI of 19.0 to 28.0 kg/m2 (including the boundary value).
* Subject have no fertility, sperm/egg donation plan for at least 6 months from the signing of the informed consent to the end of the treatment, and voluntarily takes medically recognized effective non-drug contraceptive measures (including his partner) during the trial.

Exclusion Criteria:

* Have participated in clinical trials of drugs in other trials within 3 months prior to screening .
* With clinically significant investigator-identified abnormalities of the cardiovascular, respiratory, digestive, endocrine systems (e.g., diabetes), nervous/mental systems, blood, and lymphatic systems (immune deficiency), and musculoskeletal systems.
* With clinically significant infectious disease (e.g., cellulitis, abscess, or systemic infection (e.g., sepsis), or history of clinically significant opportunistic infection (e.g.,invasive candidiasis or pneumocystis pneumonia) within 3 months before to screening.
* With a history of active tuberculosis or the presence of latent tuberculosis infection or active tuberculosis indicated by any current symptoms, signs or laboratory tests.
* Have an allergic constitution, history of allergy to the test drug ingredient or to any drug or food or pollen.
* Received chemotherapy, radiotherapy, immunosuppressive therapy, or high-dose corticosteroid treatment within 5 years before signing the informed consent.
* Use of any prescription, OTC, traditional Chinese medicine, vitamin or health product within 1 month prior to screening;
* Received live or attenuated vaccines within 1 month or have any vaccination schedule during the clinical trial.
* Had surgery within 6 months prior to screening or planned surgery during the trial.
* Have difficulty with venous blood collection, or subjects who faint at the sight of blood or a needle, or have difficulty with subcutaneous administration.
* Have lost or donated blood for more than 400 mL(not including menstrual blood loss )or received blood transfusion or using blood products within 3 months before signing informed consent or planning to donate blood during the study or within 1 month after the trial.
* Excessive consumption of tea, coffee or caffeinated beverages (more than 8 cups per day, 250 mL per cup) within 6 months prior to screening.
* Have consumed any beverage or food containing grapefruit or caffeine (such as grapefruit juice, coffee, strong tea, chocolate, caffeinated carbonated beverages, cola, cocoa, etc.) in the 48 hours prior to screening.
* Have special dietary requirements and cannot comply with a unified diet.
* Smoked ≥5 cigarettes per day within 3 months prior to screening or or could not guarantee to quit smoking during the trial.
* Regularly drank alcohol within 6 months prior to screening(i.e., more than 14 standard units per week for women and more than 21 standard units per week for men (1 standard unit containing 14g of alcohol, such as 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine) or could not abstinence during the trial; Or a positive alcohol breath test;
* With previous history of drug abuse/drug use; Or test positive for drug abuse screening (including THC, morphine, ketamine, methamphetamine, benzodiazepines, cocaine);
* Pregnant or lactating women, or positive blood pregnancy test results;
* Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV), human immunodeficiency virus (HIV) antigen-antibody combined detection, syphilis treponema specific antibody at the screening visit.
* Subjects with the results of physical examination, vital signs, laboratory examination and other auxiliary examinations (chest imaging, abdominal B-ultrasonography, 12-lead electrocardiogram, etc.) were judged by the investigator as abnormal and clinically significant during the screening period.
* The investigators considered that subjects were not suitable for this clinical trial for other reasons.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Adverse Events | up to 92 days
  incidence ,severity and relation to investigational drugs of Adverse Events according to CTCAE V5.0
Vital Signs | up to 92 days
  number of praticipants with clinically notable Vital Signs according to CTCAE V5.0
Laboratory Tests | up to 92 days
  number of praticipants with clinically notable Laboratory Tests according to CTCAE V5.0
ECG | up to 92 days
  number of praticipants with clinically notable Electrocardiogram(ECG) Values according to CTCAE V5.0
Injection Site Reaction | up to 4 days
  number of praticipants with clinically notable Injection Site Reaction according to CTCAE V5.0

SECONDARY OUTCOMES:
Pharmacokinetics-Cmax | up to 92 days
  maximum serum concentration
Pharmacokinetics-AUC 0-t | up to 92 days
  area under the concentration-time curve (AUC) from administration to the last measurable concentration
Pharmacokinetics-AUC 0-inf | up to 92 days
  AUC extrapolated to infinitymeasurable concentration
Anti-Drug antibody (ADA) | up to 92 days
  number and percentage of subjects tested ADA positive

CONTACTS AND LOCATIONS:
Overall Officials: Li J Tong, Doctor, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No